CLINICAL TRIAL: NCT01771952
Title: Prospective, Randomized, Double Blind Evaluation of the Efficacy of a Single Dose of Synvisc-One® (6.0 cc) for the Treatment of Patellofemoral Chondromalacia
Brief Title: Randomized Evaluation of the Efficacy of Synvisc-One® for the Treatment of Patellofemoral Chondromalacia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Joseph Hart, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14386
Record Dates: First submitted 2012-05-15; First posted 2013-01-18 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Chondromalacia Patella; Patellofemoral Pain Syndrome
Keywords: Patellofemoral Chondromalacia; Anterior Knee Pain; Patellofemoral Pain Syndrome; Synvisc-One; Hyaluronic Acid
MeSH Terms: conditions — Chondromalacia Patellae; Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synvisc-One™ (Experimental): Patients randomized into this group will receive a single 6cc dose of Synvisc-One™ under sterile conditions. After cutaneous numbing with vasocoolant spray, the superolateral aspect of the patellofemoral joint will be draped and prepared with betadine soaked sterile gauze using concentric circles around the injection site. A 22 gauge needle will be advanced into the patellofemoral joint using a superolateral approach. Subjects will be monitored for minimum 5 minutes post injection to evaluate for adverse events.
  Interventions: Device: Synvisc-One™
- Sham Treatment (Sham Comparator): Patients randomized into this group will receive, under sterile conditions, a sham injection. Sterile preparation and injection procedures will be exactly the same as described above except, nothing will be injected into the joint. This procedure will include a needle stick through the joint without arthrocentesis or injection.
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Device: Synvisc-One™ — A single 6cc injection of Synvisc-One™ will be utilized in this study.
  Other Names: Hyaluronan; Hyaluronic Acid
  Arms: Synvisc-One™
Other: Sham Treatment — A single needle stick without arthrocentesis or injection.
  Arms: Sham Treatment

SUMMARY:
The purpose of this study is to determine how safe a knee injection called Synvisc-One® is in patients with a condition called chondromalacia patella and how well in works in treating the condition.

Chondromalacia patella is a common cause of kneecap pain or front knee pain. Often called "Runner's Knee," this condition often affects young, otherwise healthy individuals.

Chondromalacia is due to irritation of the undersurface of the kneecap. The undersurface of the kneecap, or patella, is covered with a layer of smooth cartilage. This cartilage normally glides effortlessly across the knee during bending of the joint. In some individuals, the cartilage on the undersurface of the knee cap becomes irritated and soft, resulting in pain. Potential treatments for this condition include rest, injections (numbing or anti-inflammatory medications to reduce swelling and pain), and/or guided strengthening exercises which may help reduce pain.

Other Treatments are being evaluated. This study is about Synvisc-One® an experimental device that has been approved by the Food and Drug Administration (FDA) for the treatment of pain in osteoarthritis (OA) of the knee in patients who have failed to respond to treatments that do not involve drugs or surgery and simple pain medication such as acetaminophen. Synvisc-One® is a gel-like substance that, when injected into a joint, acts to lubricate and cushion the joint. Synvisc-One® is made from hyaluronan, which is a molecule that is found normally in joint fluid.

Synvisc-One® has not been proven to be safe or helpful in patients with chondromalacia patella (cartilage irritation or softening of the undersurface of the 'knee cap'). So far, this drug/device has been given to over 10,000 people who have knee pain (due to osteoarthritis) and has been proven safe and effective in patients with moderate to severe pain due to knee joint osteoarthritis.

DETAILED DESCRIPTION:
Study Procedures:

Screening visit:

After written informed consent is obtained, initial screening will consist of a thorough medical history and physical examination and standing, bilateral PA, lateral and merchant view x-ray evaluation. Special attention will be given to inclusion and exclusion criteria as listed above. Only patients who meet all inclusion and exclusion criteria will be allowed to continue to Baseline outcomes data collection and randomization. The following subjective outcomes, clinical examination and quadriceps strength data will be collected at each session.

Subjective Outcomes

* Knee Injury Outcome and Osteoarthritis Score (KOOS)
* Anterior knee pain rating during single-leg squat (10cm visual analog scale-VAS)

Quadriceps strength testing

• Maximal, normalized isometric knee extension force (N/kg)

Randomization:

Each subject will be randomly assigned in a 1:1 ratio to receive one of the treatments (group) described above. Randomization will be done a priori via a random number generator. Group assignments will be sealed in an envelope each containing a number from 001-100. Randomization envelope #001 will be used for the first subject, #002 for the second and so on.

Blinding:

Both examiner and patient will be blinded to treatment/ group assignment. During the injection procedure, we will block patients' view of the injection with the use of a physical screen (pillowcase, blanket, sheet, etc) in order to assure the patient is blinded to treatment. Patients will be "un-blinded" after the final study endpoints have been collected or if needed due to early withdraw or other medical emergency. To maintain blinding and avoid measurement bias, the injecting physician will be different from the investigators performing outcomes assessments.

Medication/ Treatment Restrictions and Monitoring:

* Patients will be instructed to refrain from any other intra-articular treatment or therapy while enrolled in this study
* Patients will be interviewed regarding medication usage (dosage and frequency) at each visit.
* Patients will be instructed to refrain from using any medicine for pain with the exception of OTC Tylenol.

Standardized Exercise prescription:

Patients will be prescribed a standardized home-based quadriceps strengthening program. Patients will be educated on duration and frequency for exercises and will be provided an exercise log that will provide exercise descriptions and reminders as well as a method for exercise compliance. Subjects will return exercise books at each visit for compliance recording.

Follow-up visits

* 1 month following injection: Patients will return at 4 weeks (approx 30±7 days) following injection. The following outcomes will be recorded during this visit:

  * Subjective outcomes
  * Clinical Evaluation
  * Quadriceps strength testing
  * Concomitant medications
  * Adverse Events
* 3 months following injection: Patients will return at 12 weeks (approx 91±7 days) following injection. The following outcomes will be recorded during this visit:

  * Subjective outcomes
  * Clinical Evaluation
  * Quadriceps strength testing
  * Concomitant medications
  * Adverse Events
* 6 months following injection: Patients will return at 26 weeks (approx 182±14 days) following injection. The following outcomes will be recorded during this visit:

  * Subjective outcomes
  * Clinical Evaluation
  * Quadriceps strength testing
  * Concomitant medications
  * Adverse Events

ELIGIBILITY:
Inclusion Criteria:

* Age at time of randomization: 18-45 years
* Clinical diagnosis of anterior knee pain
* X-ray showing no fracture or osteoarthritis
* >4 out of 10 on a visual analog scale and/or Knee & Osteoarthritis Outcome Score (KOOS) <7
* Persistent anterior knee pain lasting at least 3 months prior to screening
* Failed previous physical therapy intervention
* Pain/crepitus with patellar grind

Exclusion Criteria:

* Presence of knee/ patellofemoral joint effusion
* Patellar tendonitis
* Patellofemoral joint space narrowing as noted on Merchant/sunrise x-ray
* Diagnosis of tibiofemoral osteoarthritis
* Cruciate/ collateral knee ligament instability
* Patellofemoral joint instability
* Significant patellar or tibiofemoral mal-alignment
* Suspected meniscus injury
* Any clinical indication for arthroscopic surgery
* Significant patellar mal-tracking as noted on merchant view x-ray
* Currently enrolled in another experimental clinical trial
* Patellofemoral joint injection within the past 3 months
* Known or suspected psychological disorder
* Known allergy to avian products
* Oral steroid medications
* Intra-articular (knee joint) steroids in the past 6 months
* Any prior use of viscosupplements
* Pregnant or breast feeding
* Body mass index > 40
* Prior surgery in the knees (excludes debridement only procedures)
* Clinical evidence of hip disease
* Any form of inflammatory arthritis ( e.g. RA, gout, pseudogout, lupus, etc)
* Significant co-morbid conditions as determined by the investigator
* Willing to refrain from chiropractic treatment or acupuncture during the study
* Any other intra-articular knee joint injection during the study
* Kellgren Lawrence grade osteoarthritis of II, III or IV

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2010-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hart, PhD, ATC, Principal Investigator — University of Virginia; David Diduch, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Hart JM, Kuenze C, Norte G, Bodkin S, Patrie J, Denny C, Hart J, Diduch DR. Prospective, Randomized, Double-Blind Evaluation of the Efficacy of a Single-Dose Hyaluronic Acid for the Treatment of Patellofemoral Chondromalacia. Orthop J Sports Med. 2019 Jun 24;7(6):2325967119854192. doi: 10.1177/2325967119854192. eCollection 2019 Jun. PMID 31263727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synvisc-One™ | Sham Treatment
Started | 45 | 41
Completed | 42 | 38
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synvisc-One™ | Sham Treatment | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 43 | 40 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7) | 28.1 (8.4) | 27.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 45 | 41 | 86

OUTCOME MEASURES:

1. Primary Outcome: Knee Pain During a Single Leg Squat
Description: Participants will be asked to rate their worst knee pain on a visual analog scale during a deep single leg squat. The scale ranges from 0-10 where higher numbers indicate more pain. A score of 0 indicates no pain and a score of 10 indicates worst possible pain.
Time Frame: Baseline, 1 month, 3 month and 6 month
Population: 107 patients were screened, 86 were randomized (45 Synvisc one injection, 41 sham), 6 were lost to follow up leaving 42 in the Synvisc one and 38 in the sham group that completed the follow up visit and were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One™ | Sham Treatment
Number analyzed (Participants) | 45 | 41
units on a scale
  Baseline | 5.6 (1.9) | 5.2 (1.7)
  1 month: number analyzed (Participants) | 42 | 39
  1 month | 4.1 (2.5) | 3.4 (2.3)
  3 month: number analyzed (Participants) | 41 | 40
  3 month | 3.6 (2.5) | 2.2 (2.1)
  6 month: number analyzed (Participants) | 42 | 38
  6 month | 2.9 (2.4) | 2.3 (1.9)

2. Secondary Outcome: KOOS: Patient Reported Knee Function
Description: Patients will be asked to complete several validated questionnaires to assess their knee symptoms and daily function. The Knee Osteoarthritis Outcome Score (KOOS) was used as a cumulative score that included all sub-scales. The resultant score ranged from 0-100 where higher scores indicated better function.
Time Frame: Baseline, 1 month, 3 month and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Synvisc-One™ | Sham Treatment
Number analyzed (Participants) | 45 | 41
score on a scale
  Baseline | 63.5 (11.5) | 64.9 (15.5)
  1 month: number analyzed (Participants) | 42 | 39
  1 month | 68.9 (14.8) | 79.9 (11.2)
  3 month: number analyzed (Participants) | 41 | 40
  3 month | 70.7 (16.6) | 79.9 (14.9)
  6 month: number analyzed (Participants) | 42 | 38
  6 month | 74.5 (15.2) | 82.5 (11.5)

3. Secondary Outcome: Quadriceps Muscle Function
Description: Participants will contract their thigh muscle as hard as possible in order to measure their maximum strength. The outcome measure is maximum strength expressed in Newton-meters/kilogram. This outcome ranges from 0 indicating no strength to infinity where higher scores indicate stronger muscles.
Time Frame: Baseline, 1 month, 3 month and 6 month
Population: The data reported below are from 45 patients randomized to Synvisc one and 41 patients randomized to sham.
Measure: Mean (Standard Deviation); unit: Newton-meters/kilogram
Arm/Group | Synvisc-One™ | Sham Treatment
Number analyzed (Participants) | 45 | 41
Newton-meters/kilogram
  Baseline: number analyzed (Participants) | 41 | 41
  Baseline | 1.63 (.88) | 1.84 (.82)
  1 month: number analyzed (Participants) | 39 | 38
  1 month | 1.77 (.8) | 1.84 (.71)
  3 month: number analyzed (Participants) | 44 | 41
  3 month | 1.45 (.82) | 1.68 (.63)
  6 month: number analyzed (Participants) | 44 | 41
  6 month | 1.55 (.74) | 1.59 (.7)

ADVERSE EVENTS:
Arm/Group | Synvisc-One™ | Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/41
Other Adverse Events (participants affected / at risk) | 9/45 | 6/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synvisc-One™ (N=45) | Sham Treatment (N=41)
Knee pain and/or stiffness (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) — Self reported knee pain and / or knee stiffness
Knee Effusion with or without pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — Knee swelling noted on exam during research visits with or without self reported knee pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No